CLINICAL TRIAL: NCT06358547
Title: Preimplantation Genetic Testing for Aneuploidy (PGT-A) in Women Aged 37-41 Years - a Randomized Controlled Multicenter Trial
Brief Title: Preimplantation Genetic Testing for Aneuploidy (PGT-A) in Women Aged 37-41 Years
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anja Bisgaard Pinborg, Professor & medical director at the Fertility Clinic, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-23072469
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGT-A (Experimental): PGT-A and freeze-all (by vitrification) of day 5 and/or day 6 and/or day 7 blastocyst(s) and subsequent transfer of euploid or mosaic (≤80%) blastocysts in FET cycles. Luteal phase supplementation (LPS) will be administered according to the participating clinics standard practice.
  Interventions: Diagnostic Test: PGT-A
- Control (No Intervention): Non-PGT-A and fresh blastocyst transfer. In the non-PGT-A group, fresh day 5 single blastocyst transfer and/or FET of day 6 and/or day 7 blastocysts is used. LPS will be administered according to the participating clinics standard practice. All surplus day 5, day 6, or day 7 blastocysts will be vitrified. If there is a risk of OHSS, elective freeze-all will be performed. None of the blastocysts will be PGT-A tested.

INTERVENTIONS:
Diagnostic Test: PGT-A — PGT-A is a technique that allows for the prediction of embryo ploidy status through analysis of a trophectoderm biopsy conducted prior to embryo transfer.
  Arms: PGT-A

SUMMARY:
A multinational multi-centre, randomized, controlled non-blinded trial with participation of three fertility clinics in Denmark and one in Spain to assess the efficacy and safety of preimplantation genetic testing for aneuploidy (PGT-A) in 37-41-year-old women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 37-41 years with a male partner, a female partner og undergoing fertility with no partner.
* Anti Müllerian Hormone (AMH) ≥6.28 pmol/L (AMH should be measured no more than one year prior to study inclusion). The optimal is to use the Elecsys® Assay. If other assays are used this should be reported to the investigator and the AMH cut-off level may appropriately be changed so that it corresponds to the cut-off used in the Elecsys® Assay.
* IVF/ICSI cycle number 1-5 (previous IVF/ICSI cycles will not count if the woman is recruited after an IVF/ICSI/FET-delivery).

Exclusion Criteria:

* PGT-SR or PGT-M.
* Testicular sperm aspiration (TESA), testicular sperm extraction (TESE), micro-TESE (or cryopreserved sperm from these procedures).
* Males with severely compromised semen quality (<1 million progressively motile sperm cells following gradient centrifugation).
* Endometriosis stage three or four.
* Women with severe thyroid disease (women can be included if they have normal thyroid levels on relevant medication).
* Severe co-morbidity; diabetes mellitus type 1 (DM1), Mb Crohn or Colitis ulcerosa, systemic lupus erythematosus (SLE), HIV, Hepatitis B/C, or dysregulated thyroid disease.
* ≥2 previous ART treatment without blastocyst formation.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 590 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate per first embryo transfer | Approximately 12 months after inclusion of the last patient
  To assess if PGT-A is superior to standard non-PGT-A treatment regarding the live birth rate per first embryo transfer (ET) (or no ET if only aneuploid embryo(s) in the PGT-A group) per randomized woman.
Cumulative live birth rate after one complete ART treatment | Approximately 18 months after inclusion of the last patient
  To assess if PGT-A is non-inferior compared to standard treatment regarding the cumulative LBR after one complete ART treatment per randomized woman.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided